CLINICAL TRIAL: NCT05501587
Title: Measures of Respiratory Health Registry
Acronym: MRH
Status: Recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jonathan Rayment, Principle Investigator, University of British Columbia
Other Study IDs: H18-00812
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Respiratory Disease; Cystic Fibrosis
MeSH Terms: conditions — Respiration Disorders; Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Participants with CF
- Participants with other Respiratory Disease
- Healthy Participants

SUMMARY:
There are many techniques that can allow for the quantification of lung function in children; some are being used clinically and others are under development. Many of these tools are available at BC Children's Hospital. This registry study will act as a central repository for the results of traditional and novel pulmonary function tests done at BC Children's Hospital to allow for future analysis.

DETAILED DESCRIPTION:
The scope of the registry is to collect data on small airways function in healthy children, children with cystic fibrosis (CF) and children with non-CF respiratory disease using the multiple breath washout (MBW) system. These data will be stored along with demographic data, clinical data, and traditional pulmonary function testing (PFT) data. The MBW data will be collected with concurrent with clinically indicated PFT testing.

The purpose of the registry is to 1/ establish a locally collected normal range of small airways function across the paediatric age range and 2/ to collect these measurements in CF and non-CF respiratory disease.

Ultimately, the objective of this registry is to validate MBW technology as a tool that can be utilized in clinical care.

ELIGIBILITY:
Participants with CF

Inclusion Criteria:

-Diagnosis of CF as evidenced by one or more clinical feature consistent with the CF phenotype or positive CF newborn screen AND one or more of the following criteria: i. A documented sweat chloride ≥ 60 mEq/L by quantitative pilocarpine iontophoresis (QPIT).

ii. A documented genotype with two disease-causing mutations in the CFTR gene.

- In the opinion of the investigator, the participant will likely have the ability to perform the lung function test of interest on the day of testing

Exclusion Criteria:

* Physical findings at the screening that would compromise the safety of the participant or the quality of the data (e.g. respiratory distress or work of breathing)
* Requirement of supplementary oxygen to maintain oxygen saturation above 95%

Participants with other Respiratory Disease

Inclusion criteria:

* Physician-diagnosed lung disease
* Informed consent by participant, parent, or legal guardian
* In the opinion of the investigator, the participant will likely have the ability to perform the lung function test of interest on the day of testing

Exclusion criteria

* Physical findings at screening that would compromise the safety of the participant or the quality of the research data
* Requirement of supplementary oxygen to maintain oxygen saturation above 95%

Healthy Participants

* Inclusion criteria
* Informed consent by participant, parent, or legal guardian
* In the opinion of the investigator, the participant will likely have the ability to perform the lung function test of interest on the day of testing

Exclusion criteria

* Physical findings at screening that would compromise the safety of the participant or the quality of the research data
* Evidence of lung disease

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with CF Participants with other Respiratory Disease Healthy Participants
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-10-11 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
To validate new lung function testing technologies | 10 years
  The ultimate objective of this registry is to validate new lung function testing technologies as tools that can be utilized in clinical care.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Rayment, MDCM, MSc, Principal Investigator — University of British Columbia
Locations (1):
- British Columbia Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
MRH-Registry Data may be shared with investigators from BCCHR/UBC or elsewhere. MRH-Registry Co-Investigators using MRH Registry Data to address the Scientific Objectives of the MRH Registry do not need to formally apply for access. All other User-Investigators (domestic and international) must apply to the MRH-Registry Data Access Committee for access to the MRH-Registry Data.
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: Criteria for access to the MRH-Registry Data:
  The Proposed Study must demonstrate approval by a Qualified REB The objectives of the Proposed Study must align with the scientific objectives of the iMRH-Registry Use of the MRH Registry Data in the Proposed Study must respect the informed consent given by the participants of the iMRH Registry; The Proposed Study must have scientific merit, as assessed by the MRH Registry Data Access Committee The User-Investigator must demonstrate sufficient funding to perform the Proposed Study.